CLINICAL TRIAL: NCT01267188
Title: A Phase 2, Open-Label, Dose Titration Study to Evaluate the Efficacy and Safety of NBI-98854 for the Treatment of Tardive Dyskinesia in Subjects With Schizophrenia or Schizoaffective Disorder
Brief Title: Efficacy and Safety of NBI-98854 in Subjects With Tardive Dyskinesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Christopher O'Brien, MD / Chief Medical Officer, Neurocrine Biosciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-98854-1001
Record Dates: First submitted 2010-12-21; First posted 2010-12-28 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Tardive Dyskinesia
MeSH Terms: conditions — Tardive Dyskinesia | interventions — valbenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NBI-98854 (Experimental): Open-label, dose titration of active drug
  Interventions: Drug: NBI-98854

INTERVENTIONS:
Drug: NBI-98854 — powder in bottle, prepared doses at 12.5, 25, and 50 mg q.d. administered for up to 12 days consisting of three treatment periods of 4 days each

SUMMARY:
The purpose of this study is to assess the safety and efficacy of three doses (12.5, 25, and 50 mg) of NBI-98854 for the treatment of the symptoms of tardive dyskinesia (TD) in subjects with schizophrenia or schizoaffective disorder.

DETAILED DESCRIPTION:
This is a Phase 2, open-label, dose titration study to assess the efficacy and safety of three once daily (q.d.) doses (12.5, 25, and 50 mg) of NBI-98854 administered once daily for up to 12 days consisting of three treatment periods of 4 days each (Periods 1, 2, and 3). The starting dose will be 12.5 mg q.d. (Period 1), and this dose will be escalated to 25 mg q.d. (Period 2) and then to 50 mg q.d. (Period 3) based upon each subject's ability to tolerate NBI-98854. Progression to the next dose level will be based upon the subject's ability to tolerate the previous dose and the Investigator's review of adverse events and safety data. For subjects who do not tolerate a dose increase, the dose may be decreased to the dose that was previously administered (i.e., 25 mg to 12.5 mg, 50 mg to 25 mg) and continued at that dose for the remainder of the study treatment. Up to 10 medically stable subjects with schizophrenia or schizoaffective disorder who have moderate or severe symptoms of TD will be enrolled as outpatients.

ELIGIBILITY:
Inclusion Criteria:

* Males or females (non-childbearing potential) aged 18 to 65 years (both inclusive).
* Have moderate or severe Tardive Dyskinesia symptoms (Total AIMS score of at least 9)
* Have a clinical diagnosis of schizophrenia or schizoaffective disorder.
* Receiving a stable dose of antipsychotic medication for a minimum of 30 days or have stable psychiatric status.
* Doses of concurrent medications and the conditions being treated have been stable for a minimum of 30 days and expected to remain stable during the study.
* Are in good general health and expected to complete the clinical study as designed.
* Have a body mass index (BMI) of 18 to 38 kg/m^2.
* Have adequate hearing, vision, and language skills to perform the procedures specified in the protocol.

Exclusion Criteria:

* Have an active clinically significant unstable medical condition within 1 month (30 days) prior to screening.
* Have a history of substance dependence or substance (drug) or alcohol abuse within the 3 months before study start.
* Have a known history of neuroleptic malignant syndrome.
* Have a significant risk of suicidal or violent behavior.
* Receiving medication for the treatment of Tardive Dyskinesia
* Receiving any excluded concomitant medication as specified in the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Assessment of Tardive Dyskinesia symptoms | 19 days
  Abnormal Involuntary Movements Scale (AIMS) and Clinical Global Impression - Global Improvement of TD (CGI-TD) scale

SECONDARY OUTCOMES:
Number of Participants with Adverse Events following dosing with NBI-98854 | 19 days
  Outcome assessment includes monitoring of:
  * Adverse events
  * Clinical laboratory tests
  * Vital signs
  * Physical examinations
  * 12-lead electrocardiogram (ECG)
Evaluate pharmacokinetics of three doses of NBI-98854 | 19 days
  Blood samples will be collected and analyzed to evaluate drug and metabolite plasma concentrations.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto, Ontario, Canada